CLINICAL TRIAL: NCT03126474
Title: Defining Displacement Thresholds for Surgical Intervention for Distal Radius Fractures - a Delphi Study
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0593
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2017-04

CONDITIONS: Wrist Fracture; Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Delphi panel: Group of expert surgeons who have experience dealing with distal radius fractures No intervention will be performed on a patient. Participants will discuss and aim to obtain agreement about best treatment options for a variety of cases

SUMMARY:
Wrist (distal radius fractures) are very common injuries. Despite this there is still much controversy about the best way to treat them and in particular which ones require intervention. Many studies have been carried out but there is no strong evidence to answer these questions. The investigators are carrying out a Delphi study which involves seeking consensus from experts at treating these injuries about the best way to manage them. UK and international expert surgeons will take part in three rounds of online questionnaires to help decide how much displacement of the fracture will trigger treatment for different common wrist fracture cases. The aim of the study is to obtain expert opinion through consensus from the expert group about the amount of displacement that is acceptable until intervention is required.

This will provide guidance and reduce variation between treating surgeons.

DETAILED DESCRIPTION:
The investigators conducted a systematic review following SIGN guidelines with the British Society for Surgery of the Hand(BSSH) blue book committee looking at the relationship between measured radiological parameters and functional outcome. 42 studies were identified all of which were of low quality. The conclusion was; 'Currently there is insufficient evidence to demonstrate an association between any measured radiological parameters and patient rated outcome. Further high quality research is required to answer this question.' The review identified that the most commonly measured parameters were radial height, radial inclination, volar tilt and intra articular step and gap.

The Delphi process involves seeking consensus from renowned experts to provide an answer to specific research questions. Through this Delphi study the investigators intend to investigate and achieve consensus regarding the threshold for intervention in displaced distal radius fractures. The aim is to quantify how much displacement can be accepted before intervention is required for different patient groups. This can then help guide surgeons with their management decisions and help reduce variation.

A three round modified Delphi process will be used. Identified experts will be sent an invitation email with an attached electronic form which they will be asked to fill in and return to indicate if they wish to take part.

Invitation emails will be sent on the same day to all experts and they will be given 14 days to return the acceptance form.

The first round will start 14 days after the invitation email is sent. The first round electronic survey link will simultaneously be emailed to all participants who have agreed to take part. After seven days, a second e-mail (reminder) will be sent to the participants who do not respond to the first invitation. On the 15th day, responses for the first round will be collected. The investigators will analyse the collected responses and the level of agreement in the responses will be assessed.

The second round will be conducted 14 days after the first round is finalised and analysed. Only the responders who take part in the first round will be invited. The participants will be given the information about the results of the first round ,the methodology used and a review of the literature. Reminder e-mails will be sent on the 7th day, concluding the second round at 15th day. The second round results will be evaluated using the same method as that for the first round. The format of the third round (if required due to persistent disagreement) will be similar to that of the second round. Consensus is defined as 70% agreement between participants

ELIGIBILITY:
Inclusion Criteria:

* Experienced expert surgeons who regularly treat patients with distal radius fractures and/or have researched the subject extensively

Exclusion Criteria:

* Excluded if not an experienced specialist surgeon

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Experienced expert surgeons who regularly treat patients with distal radius fractures and/or have researched the subject extensively will be invited to take part. All participants will be aged over 18 years.
  The investigators defined experts in 3 ways:
  1. - experienced hand and wrist surgeons who are members of the British Society for Surgery of the Hand.
  2. - trauma surgeons who deal with these injuries and operate on them regularly.
  3. - surgeons who are also researchers who have published studies investigating outcome in patients with distal radius fractures in the last 5 years so have a comprehensive understanding of the nature of the injury and likely outcome.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2017-05-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Agreement on questions from expert panel | 10 weeks
  Agreement is defined as a consensus of 70% between expert panel members

CONTACTS AND LOCATIONS:
Overall Officials: Nick A Johnson, MBCHB, Principal Investigator — University of Leicester
Locations (1):
- Nick Johnson, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No